CLINICAL TRIAL: NCT05105178
Title: Effect of a Repeated Verbal Stimulation of Orientation on Emergence Agitation After General Anesthesia: a Randomized Double-blind Trial
Brief Title: Verbal Stimulation of Orientation on Emergence Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bo Rim Kim, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21082521254
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Emergence Delirium
Keywords: Emergence delirium, Emergence agitation, Orientation
MeSH Terms: conditions — Emergence Delirium; Orientation, Spatial

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orientation (Experimental): Information of orientation (time, place, patient's own name) is repeatedly provided during emergence.
  Interventions: Other: Giving orientation with headphones
- Name (Active Comparator): As usual, patient is recovered from general anesthesia with his/her name called.
  Interventions: Other: Emergence as usual with headphones

INTERVENTIONS:
Other: Giving orientation with headphones — During emergence, recorded voice of an investigator giving Information of orientation (time, place, patient's own name) is repeatedly played from noise-cancelling headphones
  Arms: Orientation
Other: Emergence as usual with headphones — During emergence, recorded voice of an investigator calling the patient's name is repeatedly played from noise-cancelling headphones
  Arms: Name

SUMMARY:
The purpose of this study is to investigate whether information of the orientation such as time, place, and patient's own name can reduce emergence delirium after general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic or robot-assisted abdominal surgery

Exclusion Criteria:

* Patients' refusal
* Change in operation schedule
* American Society of Anaesthesiologists (ASA) physical status Ⅳ
* Day surgery
* BMI ≥35
* Neurocognitive impairment, hearing disorder
* Psychological drug intake
* Experience of general anesthesia or sedation within 1 month

Drop out Criteria

* Changes in operation schedule (e.g. unexpected collaborative surgery, conversion to laparotomy, delay of the schedule to night-duty hours)
* Significant protocol violation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Incidence of emergence agitation at operating room (OR) | 20 minutes after anesthesia emergence
  Riker sedation agitated scale ≥5

SECONDARY OUTCOMES:
Incidence of dangerous emergence agitation | 20 minutes after anesthesia emergence
  Riker sedation agitated scale =7
maximal Riker sedation agitated scale during emergence | 20 minutes after anesthesia emergence
  maximum value of Riker sedation agitated scale during emergence
Time to emergence | 20 minutes after anesthesia emergence
  Time from anesthetics off to eye opening/extubation/discharge from OR
Bispectral index (BIS) | 20 minutes after anesthesia emergence
  BIS value at desflurane discontinuation/verbal response/extubation
Incidence of emergence agitation at PACU | 30 minutes after PACU adminstration
  Riker sedation agitated scale ≥5
Incidence of postoperative delirium | 30 minutes after PACU adminstration / Postoperative 24 hours
  Delirium scale (CAM)
Postoperative Pain | 10/20/30 minutes after PACU administation / Postoperative 24 hours
  NRS score (0-11) of pain
PACU stay | up to 3 hours after PACU administration
  Length (hours) of PACU stay
Postoperative opioid consumption | 30 minutes after PACU adminstration / Postoperative 24 hours
  Postoperative opioid requirement
Analgesics requirement | Postoperative 24 hours
  Analgesics other than opioid requirement
Postoperative quality of recovery | Postoperative 24 hours
  Korean version of quality of recovery-15

CONTACTS AND LOCATIONS:
Overall Officials: Bo Rim Kim, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee S, Sohn JY, Hwang IE, Lee HJ, Yoon S, Bahk JH, Kim BR. Effect of a repeated verbal reminder of orientation on emergence agitation after general anaesthesia for minimally invasive abdominal surgery: a randomised controlled trial. Br J Anaesth. 2023 Apr;130(4):439-445. doi: 10.1016/j.bja.2022.12.009. Epub 2023 Jan 23. PMID 36697272